CLINICAL TRIAL: NCT00000102
Title: Congenital Adrenal Hyperplasia: Calcium Channels as Therapeutic Targets
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCRR-M01RR01070-0506; M01RR001070 (NIH)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-01

CONDITIONS: Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — Nifedipine

INTERVENTIONS:
Drug: Nifedipine

SUMMARY:
This study will test the ability of extended release nifedipine (Procardia XL), a blood pressure medication, to permit a decrease in the dose of glucocorticoid medication children take to treat congenital adrenal hyperplasia (CAH).

DETAILED DESCRIPTION:
This protocol is designed to assess both acute and chronic effects of the calcium channel antagonist, nifedipine, on the hypothalamic-pituitary-adrenal axis in patients with congenital adrenal hyperplasia. The multicenter trial is composed of two phases and will involve a double-blind, placebo-controlled parallel design. The goal of Phase I is to examine the ability of nifedipine vs. placebo to decrease adrenocorticotropic hormone (ACTH) levels, as well as to begin to assess the dose-dependency of nifedipine effects. The goal of Phase II is to evaluate the long-term effects of nifedipine; that is, can attenuation of ACTH release by nifedipine permit a decrease in the dosage of glucocorticoid needed to suppress the HPA axis? Such a decrease would, in turn, reduce the deleterious effects of glucocorticoid treatment in CAH.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Congenital Adrenal Hyperplasia (CAH)
* normal ECG during baseline evaluation

Exclusion Criteria:

* history of liver disease, or elevated liver function tests
* history of cardiovascular disease

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States